CLINICAL TRIAL: NCT05654558
Title: Deep Bite Correction Using Auxiliary Intrusion Cantilevers With Initial Archwires in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mona El-Maghraby, MSc candidate, Orthodontics Department, Faculty of Dentistry, Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0049-08/2019
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Deep Overbite
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auxiliary intrusion cantilevers (Experimental): Patients received a full set of 0.022- inch slot brackets (Mini 2000, Ormco) with Roth prescription. Lower first molars received double tubed bands while 2nd molars received single bondable tubes. Leveling and alignment phase then started with 0.014 inch NiTi wires engaging all teeth and synched behind 2nd molars. Two 0.017" x 0.025" TMA (Ormco) sectional wires were attached to auxiliary tubes on 1st molars with tip back bends mesial to the molars and attached with hooks distal to lateral incisors on top of basal leveling arch wire. Amount of intrusive force was measured to range between 20 and 40 grams per side. Basal leveling arches were upgraded whenever needed. All patients were assessed after 6 months of treatment.
  Interventions: Device: Auxiliary cantilever intrusion arches on initial archwires
- Routine leveling and alignment (Active Comparator): Patients received a full set of 0.022- inch slot brackets (Mini 2000, Ormco) with Roth prescription, 1st and 2nd molars received tubes or bands according to each patient's further needs Lower arch was leveled and aligned with sequential wires starting with 14 NiTi and upgraded when needed. All patients were assessed after 6 months of treatment.
  Interventions: Device: Routine leveling and alignment

INTERVENTIONS:
Device: Auxiliary cantilever intrusion arches on initial archwires — Patients received a full set of 0.022- inch slot brackets (Mini 2000, Ormco) with Roth prescription. Lower first molars received double tubed bands while 2nd molars received single bondable tubes. Leveling and alignment phase then started with 0.014 inch NiTi wires engaging all teeth and synched behind 2nd molars. Two 0.017" x 0.025" TMA (Ormco) sectional wires were attached to auxiliary tubes on 1st molars with tip back bends mesial to the molars and attached with hooks distal to lateral incisors on top of basal leveling arch wire. Amount of intrusive force was measured to range between 20 and 40 grams per side. Basal leveling arches were upgraded whenever needed. All patients were assessed after 6 months of treatment.
  Arms: Auxiliary intrusion cantilevers
Device: Routine leveling and alignment — Patients received a full set of 0.022- inch slot brackets (Mini 2000, Ormco) with Roth prescription, 1st and 2nd molars received tubes or bands according to each patient's further needs Lower arch was leveled and aligned with sequential wires starting with 14 NiTi and upgraded when needed. All patients were assessed after 6 months of treatment.
  Other Names: Relative Intrusion
  Arms: Routine leveling and alignment

SUMMARY:
The purpose of this study was to determine the effect of auxiliary intrusion cantilevers used with resilient archwires during the leveling and alignment phase in intruding lower incisors.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition present except for third molars
* No history of previous orthodontic treatment.
* Class I or II malocclusion with minimal or no lower anterior crowding (<3 mm)
* Excessive overbite (>3 mm).

Exclusion Criteria:

* Syndromic patients as well as individuals with skeletal asymmetry
* Endodontically treated or periodontally involved loweranterior teeth.
* Need for tooth extraction in the lower arch.
* Agenesis (except for third molars)
* Any kind of tooth/root shape anomaly

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Overbite | six months
  Distance between incisal edges of upper and lower incisors measured on lateral cephalometric x-rays
True incisor intrusion | six months
  Perpendicular distance between the center of resistance of mandibular central incisor and the mandibular plane measured on lateral cephalometric x-rays
Proclination of lower incisors | six months
  Angle formed by the long axis of mandibular central incisor and mandibular plane measured on lateral cephalometric x-rays
Lower incisor intrusion and proclination | six months
  Perpendicular distance between the incisal edge of the lower central incisor and mandibular plane measured on lateral cephalometric x-rays
Lower incisor intrusion | six months
  Perpendicular distance between the apex of the lower central incisor and mandibular plane measured on lateral cephalometric x-rays
Extrusion of lower first molar | six months
  Perpendicular distance between the mesio-buccal cusp tip of the lower first molar and mandibular plane measured on lateral cephalometric x-rays
Distal tip of lower first molar | six months
  Angle formed between the long axis of lower 1st molar and mandibular plane measured on lateral cephalometric x-rays

SECONDARY OUTCOMES:
Depth of curve of Spee | six months
  Measured on dental casts by summing the right and left side maximum depths from a flat plane formed by the tips of the mandibular incisors anteriorly and the distal cusp tips of the second molars posteriorly
Depth of gingival sulcus | six months
  The sulcus depth was measured using Michigan O periodontal probe.
Width of keratinized gingiva | six months
  Measured with the aid of periodontal probe from the free gingival margin to the mucogingival junction.
Root resorption of lower incisors | six months
  Length of lower incisor roots was compared in before- and after-periapical radiographs taken with a paralleling technique.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Elmaghraby, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Hanan Ismail, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Hassan Kassem, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt